CLINICAL TRIAL: NCT05449626
Title: Validity and Reliability of Turkish Version of Bayer Activities of Daily Living Scale
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/514/227/3
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease; Activities of Daily Living
Keywords: Alzheimer's disease; Activities of Daily Living
MeSH Terms: conditions — Alzheimer Disease | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer's disease group
  Interventions: Diagnostic Test: Assessment
- Healthy Group
  Interventions: Diagnostic Test: Assessment

INTERVENTIONS:
Diagnostic Test: Assessment — The Standardized Mini-Mental Test and Clinical Dementia Rating Scale will be administered by the physician to the healthy individuals with dementia to be included in the study.

SUMMARY:
The aim of our study is to verify the validity and reliability of the Turkish version of B-GYA.

DETAILED DESCRIPTION:
Dementia refers to a condition in which individuals with brain damage have multiple cognitive deficits with impairment in activities of daily living (ADL). Therefore, the assessment of ADL is one of the main criteria for evaluating dementia. ADL disorders are often observed by caregivers before they are identified by psychometric testing, thus suggesting that ADL assessment can contribute to the early detection of dementia.

Evaluation of ADL has become increasingly important with the introduction of new drugs for Alzheimer's disease (AD), as well as being a helpful tool in diagnosis. Current guidelines have recognized the need for therapeutic intervention in AD to measure and document treatment effects on ADL. It has been emphasized that internationally validated and approved test tools to evaluate dementia are important for multinational clinical drug trials that evaluate the efficacy of anti-dementia drugs. Therefore, it is of great importance to find ADL scales that can be used internationally. Various ADL scales have been developed, such as Lawton's instrumental ADL (IADL), functional activities questionnaire (FAQ), ADCS-ADL, and Bayer ADL (B-ADL). Of these, W-ADL was developed based on an international pilot study to evaluate ADL deficits in patients from different cultural backgrounds.

Specifically, through a collaborative study conducted in four different countries during the development of the RDA, the researchers prepared 141 items and selected 25 of them that could be used internationally. The target group of the scale included elderly patients suffering from mild to moderate dementia or cognitive impairment. European countries: In the United Kingdom, Germany, and Spain, the validation study of the B-ADL was carried out in three stages. The aim of our research is to verify the validity and reliability of the Turkish version of B-ADL.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 and over
* Being literate
* Having given consent to participate in the study
* Individuals diagnosed with Alzheimer's according to the international diagnostic criteria of the American National Neurological and Communication Disorders Stroke and Alzheimer's Association (NINCDS-ADRDA) and in mild and moderate stages (<2) according to the Clinical Dementia Rating: CDR will be included in the study.

Exclusion Criteria:

* Those who did not give consent to participate in the study
* CDR>2
* Except for behavioral or functional symptoms associated with dementia, individuals with medical, psychiatric, neurological conditions, or physical disabilities that may significantly affect the performance of ADL will be excluded from the study.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 individuals and healthy individuals who were diagnosed with Alzheimer's according to the international diagnostic criteria of the American National Neurological and Communication Disorders Stroke and Alzheimer Association (NINCDS-ADRDA) and were in mild and moderate stages (<2) according to the Clinical Dementia Rating: CDR. 200 individuals found will be included
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Standardized Mini Mental Test | Up to 6 months
  For the first time, Folstein et al. [12] and found to be valid and reliable in the diagnosis of mild dementia in the Turkish population will be used. SMMT, which measures mental state, is a scale that evaluates cognitive functions in five separate sections (orientation, registration, attention and calculation, recall and language). The test can be easily applied in daily medical practice and is very suitable for screening cognitive function in the elderly. The total score is 30. The cut-off point of the scale was determined as 24.
Clinical Dementia Rating Scale | Up to 6 months
  The Clinical Dementia Rating Scale was developed by Woolf in 2016 in order to have information about the participant's memory, orientation, judgment and problem-solving ability, functionality outside the home, home life, hobbies and personal care. An evaluation will be made by asking detailed questions about all the areas specified in this test, which will be applied to the patient and their relatives. According to the answers given in each field, it will be scored as 0-0.5-1-2-3 by using the score table in the front of the test. It is a general assessment made to determine the dementia stage of the person. 0.5-1 mild, 1-2 moderate, 2-3 advanced stages of dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided